CLINICAL TRIAL: NCT00647543
Title: A Multicenter, Eight-Week Treatment, Single-Step Titration, Open-Label Study Assessing The Percentage Of Dyslipidemic Patients Achieving LDL Cholesterol Target With Atorvastatin Starting Doses Of 10 Mg, 20 Mg, And 40 Mg
Brief Title: Atorvastatin Study For The Treatment Of High Cholesterol In Patients From Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2581111
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Risk (Experimental)
  Interventions: Drug: Atorvastatin
- Low Risk (Experimental)
  Interventions: Drug: Atorvastatin
- Medium Risk (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin tablets at starting doses of 10, 20, or 40 mg once daily for at least 8 weeks. Patients who achieved their LDL-C target by Week 4 continued on their starting dose for the next 4 weeks. Patients who did not achieve their LDL-C target by Week 4 were titrated up 1 dose step for the next 4 weeks.
  Arms: High Risk
Drug: Atorvastatin — Atorvastatin tablets at starting doses of 10, 20, or 40 mg once daily for at least 8 weeks. Patients who achieved their LDL-C target by Week 4 continued on their starting dose for the next 4 weeks. Patients who did not achieve their LDL-C target by Week 4 were titrated up 1 dose step for the next 4 weeks.
  Arms: Low Risk
Drug: Atorvastatin — Atorvastatin tablets at starting doses of 10, 20, or 40 mg once daily for at least 8 weeks. Patients who achieved their LDL-C target by Week 4 continued on their starting dose for the next 4 weeks. Patients who did not achieve their LDL-C target by Week 4 were titrated up 1 dose step for the next 4 weeks.
  Arms: Medium Risk

SUMMARY:
The purpose of this study is to evaluate the efficacy of atorvastatin in lowering cholesterol on patients from Thailand with high cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Dyslipidemic patients who were eligible for lipid lowering therapy
* Willingness to follow study diet for 1 month prior to screening and for the duration of the study

Exclusion Criteria:

* Use of other lipid lowering agents (6-week washout period)
* Uncontrolled high blood pressure
* Impaired liver function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2003-08; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who achieved low-density lipoprotein cholesterol (LDL-C) target | Week 8

SECONDARY OUTCOMES:
Adverse events and laboratory test changes | Weeks 2, 4, and 8
Percentage of patients who achieved LDL-C target | Weeks 2 and 4, and Week 8 with 1 step titration
Change and percent change from baseline in LDL-C | Weeks 2, 4, and 8
Change and percent change from baseline in high-density lipoprotein cholesterol (HDL-C) | Weeks 2, 4, and 8
Change and percent change from baseline in LDL/HDL ratio | Weeks 2, 4, and 8
Change and percent change from baseline in total cholesterol | Weeks 2, 4, and 8
Change and percent change from baseline in triglycerides | Weeks 2, 4, and 8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Thailand (2):
  - Pfizer Investigational Site, Bangkok
  - Pfizer Investigational Site, Chiang Mai
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581111&StudyName=Lipitor%20Study%20For%20The%20Treatment%20Of%20High%20Cholesterol%20In%20Patients%20From%20Thailand